CLINICAL TRIAL: NCT06090305
Title: Effectiveness of a Digital Health Application for Multiple Sclerosis (Levidex): Randomized Controlled Trial
Brief Title: Effectiveness of a Digital Health Application for Multiple Sclerosis (Levidex)
Acronym: LAMONT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: University Hospital Schleswig-Holstein (Other); Universität Duisburg-Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: levidex RCT 2023
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants allocated to the intervention group will receive access to levidex in addition to treatment as usual (TAU). levidex is a digital health application designed for individuals with Multiple Sclerosis (MS), accessible through a web browser. The application comprises 16 modules, with the majority focusing on treatment methods derived from cognitive behavioral therapy (CBT) and health behavior change. The program operates through interactive "dialogues", which are accompanied by illustrations, audio recordings, motivating text messages, worksheets, and summaries. Users are also encouraged to regularly complete short questionnaires to monitor their complaints. Once registered, the program remains accessible for 365 days.
  Interventions: Behavioral: levidex; Other: treatment as usual (TAU)
- Control group (Active Comparator): Participants allocated to the control group will receive an overview of relevant brochures from the Deutsche Multiple Sklerose Gesellschaft (German Multiple Sclerosis Society) on the topic of lifestyle in Multiple Sclerosis (MS) in addition to treatment as usual (TAU). After 6 months, they will be offered access to levidex.
  Interventions: Behavioral: Control; Other: treatment as usual (TAU)

INTERVENTIONS:
Behavioral: levidex — Participants will receive access to the digital health application levidex in addition to treatment as usual (TAU).
  Arms: Intervention group
Behavioral: Control — Participants will receive access to an overview of relevant brochures from the Deutsche Multiple Sklerose Gesellschaft (German Multiple Sclerosis Society) on the topic of lifestyle in MS in addition to treatment as usual (TAU).
  Arms: Control group
Other: treatment as usual (TAU) — treatment as usual (TAU)

SUMMARY:
The trial aims to evaluate the effectiveness of a novel digital health application (levidex), which was designed to increase quality of life in persons with multiple sclerosis (MS). Therefore, 470 people with MS will be recruited and randomized to two groups: (1) an intervention group that will receive access to levidex in addition to treatment as usual (TAU) (n = 235) and (2) a control group receiving an overview of relevant brochures from the Deutsche Multiple Sklerose Gesellschaft (German Multiple Sclerosis Society) on the topic of lifestyle in MS in addition to TAU (n = 235).The primary outcome measure is the total score on the Hamburg Quality of Life Questionnaire for Multiple Sclerosis (HALEMS), collected 6 months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Impaired health-related quality of life (total score of the Hamburg Quality of Life Questionnaire for Multiple Sclerosis [HALEMS] ≥ 2)
* Specialist treatment in the last three months before study inclusion
* Diagnosis of MS (relevant ICD-10-GM diagnoses G35.x), confirmed by a medical document or equivalent certificate
* Sufficient cognitive and motor skills to use an online program
* Consent to participate
* Sufficient knowledge of the German language
* Access to the Internet

Exclusion Criteria:

* Presence of severe impairment of independence or abilities (degree of care ["Pflegegrad", § 15 SGB XI] ≥ 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Hamburg Quality of Life Questionnaire for Multiple Sclerosis (HALEMS) | 6 months after randomization
  The HALEMS measures MS-specific quality of life. It covers the following domains: fatigue, thinking, mobility lower limb, mobility upper limb, communication and mood. The total score is calculated as the average of the scores in the six domains and ranges from 1 to 5. Higher scores represent lower quality of life.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 3 and 6 months after randomization
  The PHQ-9 measures depressive symptoms. Each of the 9 items is answered on a 4-point Likert scale ranging from 0 (not at all) to 3 (almost every day). The total score ranges from 0 to 27. Higher scores represent higher depressive symptoms.
Work and Social Assessment Scale (WSAS) | 3 and 6 months after randomization
  The WSAS measures an individual's perception of work and social functioning. It consists of 5 items that are answered on a 9-point Likert scale ranging from 0 (not at all impaired) to 8 (very severely impaired). The total score has a range of 0-40, with higher scores representing higher disability.
Global index score of the Multiple Sclerosis International Quality of Life (MuSiQoL) | 3 and 6 months after randomization
  The MuSiQoL measures MS-specific quality of life. It comprises 31 items covering 9 domains (activities of daily living, psychological well-being, symptoms, relationships with friends, relationships with family, relationships with the healthcare system, sentimental and sexual life, coping, and rejection). Each item is scored on a 6-point Likert scale. The score on each dimension is obtained by computing the mean of the item scores for that dimension. All dimension scores are linearly transformed to a 0-100 scale. The global index score is computed as the mean of the dimension scores. Higher scores represent higher quality of life.
Generalized Anxiety Disorder Scale-7 (GAD-7) | 3 and 6 months after randomization
  The GAD-7 is a 7-item self-report anxiety questionnaire. Items are rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). The total score can range from 0 to 21, higher scores representing higher anxiety.
Frenchay Activities Index (FAI) | 3 and 6 months after randomization
  The FAI assesses participation in social and lifestyle activities with 15 items that are scored on a 4-point Likert scale ranging from 1 to 4. It covers three subdomains (domestic chores, outdoor, work/leisure activities). The total score ranges from 15 to 60. Higher scores represent more activity.
Hamburg Quality of Life Questionnaire for Multiple Sclerosis (HALEMS) | 3 months after randomization
  The HALEMS measures MS-specific quality of life. It covers the following domains: fatigue, thinking, mobility lower limb, mobility upper limb, communication and mood. The total score is calculated as the average of the scores in the six domains and ranges from 1 to 5. Higher scores represent lower quality of life.

OTHER OUTCOMES:
HALEMS Subscales (cognition; fatigue; mobility lower limb; mobility upper limb; communication; and mood) | 3 and 6 months after randomization
  The HALEMS measures MS-specific quality of life. It covers the following domains: fatigue, thinking, mobility lower limb, mobility upper limb, communication and mood. each domain score ranges from 1 to 5. Higher scores represent lower quality of life.
Intake of disease-modifying drugs overall (last 3 months) | 3 and 6 months after randomization
Intake of DMDs classified according to efficacy (category 1-3, according to current German clinical guideline) (last 3 months) | 3 and 6 months after randomization
Number of days on sick leave/sick pay (last 3 months) | 3 and 6 months after randomization
Number of days in inpatient treatment (last 3 months) | 3 and 6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Jauch-Chara, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- GAIA AG, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No